CLINICAL TRIAL: NCT00926900
Title: The Role of the Glutamatergic System in the Extinction of Conditioned Reinforcement Processes
Acronym: SFB636D6
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Institute of Mental Health, Mannheim (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SFB636 D6 2006-007090-72
Record Dates: First submitted 2009-06-22; First posted 2009-06-24 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Alcohol Drinking
Keywords: Alcoholism; D-cycloserine; extinction; cue-exposure
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Cycloserine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D-cycloserine (Active Comparator)
  Interventions: Drug: D-cycloserine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cycloserine — 50 mg at approximately 1.5 hours prior to cue-exposure training sessions
  Arms: D-cycloserine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of this project is to explore whether the extinction of cue-reactivity following a cue-exposure based intervention in volunteers with an alcohol dependence is facilitated by drugs that increase NMDA-receptor function.

It is hypothesised that targeted treatment with D-Cycloserine prior to each extinction training session enhances the effects on cue-reactivity.

Further, a significant correlation between the reduction of cue-reactivity and both reduced craving and relapse probability is expected.

ELIGIBILITY:
Inclusion Criteria:

* current DSM-IV/ ICD-10 diagnosis of alcohol dependence
* controlled abstinence for a period of 5 to 21 days following admission to inpatient detoxification or day-clinic care
* women (in childbearing age): use of a highly effective method of contraception
* normal or corrected-to-normal vision
* ability to provide written informed consent

Exclusion Criteria:

* diagnosis of additional axis I or II disorders (according to DSM-IV( ICD- 10 criteria) either currently or within the past 12 months (except nicotine dependence)
* positive drug screening
* current medication with anti-convulsive or psychotropic drugs
* MRI ineligibility
* sensitivity to study medication as evidenced by a history of adverse drug experience
* severe withdrawal symptoms (e.g. convulsions, delirium)
* disposition towards experiencing convulsions/ epilepsy
* history of schizophrenic disorders/ affective psychosis
* neurological diseases that might affect the dopaminergic, limbic and frontal cortices or extrapyramidal motor functioning
* major diseases (e.g. diabetes, liver cirrhosis, heart disease)
* physical illness interfering with study procedures or affecting study outcomes
* pregnancy (positive test results)/ lactation period
* suicidal tendencies/ increased risk that others might be harmed -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
reduction in cue-reactivity to alcohol-associated stimuli assessed by functional magnetic resonance imaging | following completion of cue-exposure therapy

SECONDARY OUTCOMES:
time to first severe relapse to alcohol consumption | at 3 and 6 months after treatment completion

CONTACTS AND LOCATIONS:
Overall Officials: Falk Kiefer, Professor, Principal Investigator — Central Institute of Mental Health, Department of Addictive Behavior and Addiction Medicine
Locations (1):
- Central Institute of Mental Health, Mannheim, Germany

REFERENCES:
- [Derived] Strosche A, Zhang X, Kirsch M, Hermann D, Ende G, Kiefer F, Vollstadt-Klein S. Investigation of brain functional connectivity to assess cognitive control over cue-processing in Alcohol Use Disorder. Addict Biol. 2021 Jan;26(1):e12863. doi: 10.1111/adb.12863. Epub 2020 Jan 6. PMID 31908107
- [Derived] Vollstadt-Klein S, Loeber S, Kirsch M, Bach P, Richter A, Buhler M, von der Goltz C, Hermann D, Mann K, Kiefer F. Effects of cue-exposure treatment on neural cue reactivity in alcohol dependence: a randomized trial. Biol Psychiatry. 2011 Jun 1;69(11):1060-6. doi: 10.1016/j.biopsych.2010.12.016. Epub 2011 Feb 3. PMID 21292243